CLINICAL TRIAL: NCT07078721
Title: Efficacy and Safety Study of Umbilical Cord Blood Transplantation (UCBT) With Total Marrow Irradiation (TMI)-Based Conditioning Regimen for Adults With Refractory/Relapsed Aplastic Anemia (AA).
Brief Title: Efficacy and Safety of UCBT With TMI -Based Conditioning Regimen for Adults With Refractory/Relapsed Aplastic Anemia
Acronym: TMI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, SunZimin, Principal Investigator, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025071
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Aplastic Anemia Idiopathic
Keywords: aplastic anemia; refractory/relapsed; Total Marrow Irradiation; Umbilical Cord Blood Transplantation
MeSH Terms: conditions — Anemia, Aplastic; Recurrence | interventions — fludarabine; Melphalan; Honey

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TMI in AA (Experimental): Efficacy and Safety Study of Umbilical Cord Blood Transplantation (UCBT) with Total Marrow Irradiation (TMI)-Based Conditioning Regimen for Adults with Refractory/Relapsed Aplastic Anemia (AA)
  Interventions: Radiation: Total Marrow Irradiation; Drug: Fludarabine (FLU); Drug: Melphalan (Mel)

INTERVENTIONS:
Radiation: Total Marrow Irradiation — - TMI 4 Gy qd on Day -2;
  Other Names: Marrow-Targeted Radiotherapy; Organ-Sparing Marrow-Targeted Irradiation (OSMI)
Drug: Fludarabine (FLU) — Flu 30 mg/m² × 5 days on Days -6, -5, -4, -3, -2;
  Other Names: FaraA
Drug: Melphalan (Mel) — Mel 100 mg/m² qd on Day -1.
  Other Names: L-PAM

SUMMARY:
Refractory/relapsed aplastic anemia (AA) in adults remains a clinical challenge that is frequently encountered and urgently needs to be resolved. Salvage treatment should prioritize hematopoietic stem cell transplantation (HSCT). Unrelated cord blood is an ideal source of hematopoietic stem cells due to its easy availability, low immunogenicity, and low incidence of chronic graft-versus-host disease (cGVHD) after transplantation.The optimization of the conditioning regimen for UCBT is a crucial factor in determining patient outcomes.

This is a Phase II clinical study. A total of 11 adult patients with refractory/relapsed AA will be treated with a UCBT regimen based on a TMI-based conditioning regimen. Patients who meet the inclusion/exclusion criteria will sign an informed consent form before undergoing cord blood transplantation. The efficacy (12-month EFS) and safety of the regimen will be assessed 12 months after transplantation.

DETAILED DESCRIPTION:
Refractory/relapsed aplastic anemia (AA) in adults remains a clinical challenge that is frequently encountered and urgently needs to be resolved. Refractory AA is ineffective to the standard first-line treatment regimen, which is based on antithymocyte globulin (ATG) combined with cyclosporine A (CsA) as the standard immunosuppressive therapy (IST), accounting for approximately 30%-40% of all AA patients. It has been reported that the 5-year mortality rate of refractory severe aplastic anemia (r-SAA) exceeds 40% after diagnosis. Brosdky et al. reported that the 10-year event-free survival (EFS) of SAA treated with high-dose cyclophosphamide-based IST is only 28%. The efficacy is not satisfactory. Thrombopoietin receptor agonists such as eltrombopag, as an important treatment for r-SAA, have a hematologic response rate of only 41.8% with monotherapy for 52 weeks, with an overall low response rate and unsatisfactory quality of response. The 24-week complete blood count response is only 16.4%, and the 52-week response is only 21.8%. Clonal hematopoiesis is also a long-term concern for IST. Multiple centers have reported that the early efficacy of IST combined with thrombopoietin receptor agonists for treating SAA has improved, but the long-term overall efficacy has not substantially exceeded that of IST alone. The bone marrow failure of non-severe aplastic anemia (NSAA) is less severe than that of SAA, and the main treatment methods are IST ± thrombopoietin receptor agonists or combined with androgens, similar to SAA, with similar long-term efficacy challenges. Therefore, the development of new and effective treatment methods is an urgent clinical need.

Refractory AA is ineffective to IST, possibly mainly due to the insufficient number or functional abnormalities of residual hematopoietic stem/progenitor cells in patients. Therefore, salvage treatment should prioritize hematopoietic stem cell transplantation (HSCT) to supplement normal hematopoietic stem cells and rebuild hematopoiesis. According to domestic and international guidelines for the diagnosis and treatment of adult AA, unrelated donor allogeneic hematopoietic stem cell transplantation or haploidentical hematopoietic stem cell transplantation are the main salvage treatment methods for refractory SAA, with hematopoietic stem cells mainly derived from peripheral blood or bone marrow. However, the availability of suitable donors is one of the main difficulties for unrelated donor allogeneic hematopoietic stem cell transplantation or haploidentical hematopoietic stem cell transplantation. Many AA patients cannot receive early treatment due to the lack of suitable hematopoietic stem cell donors and have to wait for a long time. Unrelated cord blood is an ideal source of hematopoietic stem cells due to its easy availability, low immunogenicity, and low incidence of chronic graft-versus-host disease (cGVHD) after transplantation. However, Delatour et al. reported that the 3-year overall survival (OS) of patients with refractory AA treated with cord blood transplantation is only 38% ± 6%, with unsatisfactory efficacy. Nevertheless, with the optimization of conditioning regimens, the popularization of high-resolution HLA typing, and the continuous improvement of supportive care, the efficacy of unrelated cord blood transplantation (UCBT) is expected to improve.

The optimization of the conditioning regimen for UCBT is a crucial factor in determining patient outcomes. Hiramoto et al. reported that patients received conditioning regimens of total body irradiation (TBI) (≤4Gy) combined with fludarabine/melphalan (Flu/Mel) or fludarabine/cyclophosphamide (Flu/Cy). The results showed that a radiation dose of 4 Gy is an independent influencing factor for neutrophil engraftment. Compared with the Flu/Cy group, a higher proportion of patients in the Flu/Mel group received 4 Gy (96% vs. 68%, p<0.01), but there was no difference in engraftment success rates (77.8% vs. 72%). Compared with TBI, TMI has many advantages: (1) TMI clears residual T cells in the recipient's body, optimizes spatial competition, and better prepares the bone marrow niche for cord blood stem cells; (2) It can more accurately target the bone marrow region; (3) It reduces toxicity to other organs and can better protect the patient's organ function; (4) It reduces the risk of long-term tumors; (5) It lowers the radiation dose: the TMI dose is 4-6 Gy, while the TBI dose reaches 12 Gy; (6) TMI is applicable to a wider range of people and is more tolerable for elderly/weak patients. Therefore, TMI has potential advantages in the conditioning regimen for refractory/relapsed severe aplastic anemia.

Therefore, we have designed and proposed for the first time the Phase II clinical study titled "A Phase II Study on the Efficacy and Safety of Umbilical Cord Blood Transplantation (UCBT) with a Total Marrow Irradiation (TMI)-Based Conditioning Regimen for the Treatment of Refractory/Relapsed Aplastic Anemia (AA) in Adults." This study employs a TMI (4 Gy)/Flu/Mel conditioning regimen and single-unit cord blood stem cell transplantation to treat adult refractory/relapsed AA, aiming to evaluate the efficacy and safety of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suitable for enrollment in this study must meet all of the following criteria:

  1. Age ≥18 years and <50 years, regardless of gender.
  2. Diagnosis of AA according to the guidelines of the British Society for Haematology. The bone marrow shows hypocellularity, without infiltration of abnormal cells or marrow fibrosis. The peripheral blood must meet at least two of the following three criteria: absolute neutrophil count (ANC) <1.5×10⁹/L; platelet count <50×10⁹/L; hemoglobin <100 g/L. Based on the severity of the disease, AA is classified into severe aplastic anemia (SAA) and non-severe aplastic anemia (NSAA).

     The diagnostic criteria for severe aplastic anemia (SAA) are as follows:

     Peripheral blood criteria

     At least two of the following three criteria must be met:

     Absolute neutrophil count (ANC) <0.5×10⁹/L; Reticulocyte count <20×10⁹/L; Platelet count <20×10⁹/L; Bone marrow criteria The degree of bone marrow cellularity is <25% of normal; if ≥25% but <50% of normal, then the proportion of residual hematopoietic cells should be <30%.

     Bone marrow aspiration results show hypocellular or severely hypocellular marrow, with a marked decrease in hematopoietic cells and an increase in non-hematopoietic cells such as lymphocytes and reticular cells.

     Other：Other diseases causing pancytopenia, such as myelodysplastic syndrome (MDS), paroxysmal nocturnal hemoglobinuria (PNH), and congenital marrow failure syndromes, should be excluded.

     If ANC <0.2×10⁹/L, the diagnosis is very severe aplastic anemia (VSAA); Those who do not meet the criteria for SAA are classified as non-severe aplastic anemia (NSAA);
  3. Meet the criteria for refractory AA: ①SAA: no response to first-line ATG + CSA treatment for more than 6 months; ②NSAA: ①persistent transfusion dependence of two or more blood cell lines, ②meet any of the following criteria: no response to immunosuppressive therapy with cyclosporine for more than 12 months, or no response to androgen and/or TPO receptor agonist therapy for more than 6 months, ④or progression to SAA; Meet the criteria for relapsed AA: initially effective to first-line immunosuppressive therapy, but pancytopenia recurs after reduction or discontinuation of immunosuppressive therapy, meeting the criteria for SAA.
  4. Karnofsky score ≥60, ECOG score ≤2, HCT-CI index ≤2.
  5. No HLA-identical sibling donor or no HLA-identical unrelated donor available.
  6. Understanding of the study procedures and voluntary written informed consent.

Exclusion Criteria:

* Subjects with any of the following conditions are not eligible for enrollment in this study:

  1. Pancytopenia and hypoplastic marrow diseases caused by other reasons (including PNH, etc.).
  2. Use of intermediate or high doses of cyclophosphamide (≥20mg/kg/d) for immunosuppressive therapy within 3 months before enrollment.
  3. History of hematopoietic stem cell transplantation.
  4. Known or suspected contraindications or allergies to fludarabine, melphalan, or other drugs.
  5. Patients with uncontrolled bleeding and/or infection after standard treatment before screening.
  6. Active viral hepatitis (hepatitis B, hepatitis C, etc.), HIV infection, or syphilis at baseline or screening.
  7. Creatinine clearance rate <60 ml/min before treatment, or serum creatinine >140 μmol/L.
  8. Pregnant or breastfeeding women.
  9. Participation in another clinical trial within 3 months before enrollment.
  10. Any other condition that the investigator deems may prevent the subject from completing the study or pose significant risks to the subject.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) at 12 months post-transplant. | ---Enrollment Period (2 weeks)---Treatment Period (7 days)---Follow-Up Period (12 months)
  Event-free survival (EFS): Defined as the time from the start of UCBT to the occurrence of an event, including death, graft failure, lack of response, relapse, and clonal progression.

CONTACTS AND LOCATIONS:
Overall Officials: Zimin Sun, Principal Investigator — IH & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, City, China

IPD SHARING:
Plan to Share IPD: Yes
This is a Phase II clinical study. A total of 11 adult patients with refractory/relapsed AA will be treated with a UCBT regimen based on a TMI-based conditioning regimen. Patients who meet the inclusion/exclusion criteria will sign an informed consent form before undergoing cord blood transplantation. The efficacy (12-month EFS) and safety of the regimen will be assessed 12 months after transplantation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: start date: June 2028 end date: june 2030
Access Criteria: the users of "ClinicalTrail.gov"
URL: https://clinicaltrials.gov/

REFERENCES:
- [Background] Olnes MJ, Scheinberg P, Calvo KR, Desmond R, Tang Y, Dumitriu B, Parikh AR, Soto S, Biancotto A, Feng X, Lozier J, Wu CO, Young NS, Dunbar CE. Eltrombopag and improved hematopoiesis in refractory aplastic anemia. N Engl J Med. 2012 Jul 5;367(1):11-9. doi: 10.1056/NEJMoa1200931. PMID 22762314
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383
- [Background] Harris AC, Young R, Devine S, Hogan WJ, Ayuk F, Bunworasate U, Chanswangphuwana C, Efebera YA, Holler E, Litzow M, Ordemann R, Qayed M, Renteria AS, Reshef R, Wolfl M, Chen YB, Goldstein S, Jagasia M, Locatelli F, Mielke S, Porter D, Schechter T, Shekhovtsova Z, Ferrara JL, Levine JE. International, Multicenter Standardization of Acute Graft-versus-Host Disease Clinical Data Collection: A Report from the Mount Sinai Acute GVHD International Consortium. Biol Blood Marrow Transplant. 2016 Jan;22(1):4-10. doi: 10.1016/j.bbmt.2015.09.001. Epub 2015 Sep 16. PMID 26386318
- [Background] Kurtzberg J, Troy JD, Page KM, El Ayoubi HR, Volt F, Maria Scigliuolo G, Cappelli B, Rocha V, Ruggeri A, Gluckman E. Unrelated Donor Cord Blood Transplantation in Children: Lessons Learned Over 3 Decades. Stem Cells Transl Med. 2023 Jan 30;12(1):26-38. doi: 10.1093/stcltm/szac079. PMID 36718114
- [Background] Hiramoto N, Yamazaki H, Nakamura Y, Uchida N, Murata M, Kondo T, Yoshioka S, Eto T, Nishikawa A, Kimura T, Ichinohe T, Atsuta Y, Onishi Y, Suzuki R, Mori T; Adult Aplastic Anemia Working Group of the Japanese Society for Hematopoietic Cell Transplantation. Total body irradiation-containing conditioning regimens without antithymocyte globulin in adults with aplastic anemia undergoing umbilical cord blood transplantation. Ann Hematol. 2022 Jan;101(1):165-175. doi: 10.1007/s00277-021-04664-z. Epub 2021 Sep 21. PMID 34546409
- [Background] Peffault de Latour R, Purtill D, Ruggeri A, Sanz G, Michel G, Gandemer V, Maury S, Kurtzberg J, Bonfim C, Aljurf M, Gluckman E, Socie G, Passweg J, Rocha V. Influence of nucleated cell dose on overall survival of unrelated cord blood transplantation for patients with severe acquired aplastic anemia: a study by eurocord and the aplastic anemia working party of the European group for blood and marrow transplantation. Biol Blood Marrow Transplant. 2011 Jan;17(1):78-85. doi: 10.1016/j.bbmt.2010.06.011. Epub 2010 Jun 16. PMID 20561593
- [Background] Red Blood Cell Disease (Anemia) Group, Chinese Society of Hematology, Chinese Medical Association. [Guidelines for the diagnosis and management of aplastic anemia in China (2022)]. Zhonghua Xue Ye Xue Za Zhi. 2022 Nov 14;43(11):881-888. doi: 10.3760/cma.j.issn.0253-2727.2022.11.001. No abstract available. Chinese. PMID 36709177
- [Background] Valdez JM, Scheinberg P, Nunez O, Wu CO, Young NS, Walsh TJ. Decreased infection-related mortality and improved survival in severe aplastic anemia in the past two decades. Clin Infect Dis. 2011 Mar 15;52(6):726-35. doi: 10.1093/cid/ciq245. PMID 21367725
- [Background] Peffault de Latour R, Kulasekararaj A, Iacobelli S, Terwel SR, Cook R, Griffin M, Halkes CJM, Recher C, Barraco F, Forcade E, Vallejo JC, Drexler B, Mear JB, Smith AE, Angelucci E, Raymakers RAP, de Groot MR, Daguindau E, Nur E, Barcellini W, Russell NH, Terriou L, Iori AP, La Rocca U, Sureda A, Sanchez-Ortega I, Xicoy B, Jarque I, Cavenagh J, Sicre de Fontbrune F, Marotta S, Munir T, Tjon JML, Tavitian S, Praire A, Clement L, Rabian F, Marano L, Hill A, Palmisani E, Muus P, Cacace F, Frieri C, van Lint MT, Passweg JR, Marsh JCW, Socie G, Mufti GJ, Dufour C, Risitano AM; Severe Aplastic Anemia Working Party of the European Society for Blood and Marrow Transplantation. Eltrombopag Added to Immunosuppression in Severe Aplastic Anemia. N Engl J Med. 2022 Jan 6;386(1):11-23. doi: 10.1056/NEJMoa2109965. PMID 34986284
- [Background] Kulasekararaj A, Cavenagh J, Dokal I, Foukaneli T, Gandhi S, Garg M, Griffin M, Hillmen P, Ireland R, Killick S, Mansour S, Mufti G, Potter V, Snowden J, Stanworth S, Zuha R, Marsh J; BSH Committee. Guidelines for the diagnosis and management of adult aplastic anaemia: A British Society for Haematology Guideline. Br J Haematol. 2024 Mar;204(3):784-804. doi: 10.1111/bjh.19236. Epub 2024 Jan 21. PMID 38247114
- See also: Efficacy and Safety Study of Umbilical Cord Blood Transplantation (UCBT) with Total Marrow Irradiation (TMI)-Based Conditioning Regimen for Adults with Refractory/Relapsed Aplastic Anemia (AA) — https://clinicaltrials.gov/
- Available data/document: Study Protocol: TMI in AA — https://clinicaltrials.gov/ — Efficacy and Safety Study of Umbilical Cord Blood Transplantation (UCBT) with Total Marrow Irradiation (TMI)-Based Conditioning Regimen for Adults with Refractory/Relapsed Aplastic Anemia (AA)
- Available data/document: Informed Consent Form: TMI in AA — https://clinicaltrials.gov/ — Efficacy and Safety Study of Umbilical Cord Blood Transplantation (UCBT) with Total Marrow Irradiation (TMI)-Based Conditioning Regimen for Adults with Refractory/Relapsed Aplastic Anemia (AA)
- Available data/document: Clinical Study Report: TMI in AA — https://clinicaltrials.gov/ — Efficacy and Safety Study of Umbilical Cord Blood Transplantation (UCBT) with Total Marrow Irradiation (TMI)-Based Conditioning Regimen for Adults with Refractory/Relapsed Aplastic Anemia (AA)

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT07078721/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT07078721/ICF_001.pdf